CLINICAL TRIAL: NCT04184115
Title: A Randomized, Double Blind, Placebo-Controlled Phase 3 Study of the Safety, Efficacy and Pharmacokinetics of DPI-386 Nasal Gel for the Prevention and Treatment of Nausea Associated With Motion Sickness
Brief Title: Nasal Gel for the Prevention and Treatment of Nausea Associated With Motion Sickness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPI-386-MS-22
Record Dates: First submitted 2019-06-06; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: study is double-blinded placebo controlled for all treatment arms. All DPI-386 Nasal Gel and placebo nasal gel vials are opaque and indistinguishable. The DPI-386 Nasal Gel and placebo nasal gels are identical in color and viscosity, and without identifiable smell. Each placebo patch is similar in color and size as the TDS patch but does not deliver any medication or contain any excipients. A designated independent (unblinded) applicator will administer all patch application and removal, including an opaque waterproof bandage cover over the patch, to further prevent unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DPI-386 Nasal Gel + placebo patch (Experimental): DPI-386 Nasal Gel: Each 0.12 gram of the gel contains 0.2 mg of scopolamine HBr
  Interventions: Drug: DPI-386 Nasal Gel; Drug: Placebos
- Placebo nasal gel + Placebo patch (Placebo Comparator): Placebo
  Interventions: Drug: Placebos
- placebo nasal gel + TDS patch (Active Comparator): Transderm Scop® is a commercial transdermal scopolamine (TDS) patch worn behind the ear containing a 1.5 mg reservoir of scopolamine to be delivered over a 72-hour period.
  Interventions: Drug: DPI-386 Nasal Gel; Drug: Placebos

INTERVENTIONS:
Drug: DPI-386 Nasal Gel — 1.5 mg reservoir of scopolamine to be delivered over a 72-hour period
  Other Names: Transderm Scop®
  Arms: DPI-386 Nasal Gel + placebo patch; placebo nasal gel + TDS patch
Drug: Placebos — Placebo Nasal Gel and placebo patch

SUMMARY:
Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study to identify the safety, efficacy and pharmacokinetics of a repeated-dose regimen of DPI 386 nasal gel (intranasal scopolamine gel) for the prevention and treatment of nausea associated with motion sickness.

DETAILED DESCRIPTION:
This Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study to identify the safety, efficacy and pharmacokinetics of a repeated-dose regimen of DPI 386 nasal gel (intranasal scopolamine gel) for the prevention and treatment of nausea associated with motion sickness. The study will have three arms: DPI-386 nasal gel, placebo nasal gel, and TDS patch (1.5 mg/72 hours), the current standard of care for the treatment of motion sickness. The study will include 34 subjects per arm, for a total of 102 subjects (n=102). A double dummy design will be used to mask the treatment assignment. All subjects will receive both a patch and nasal gel randomized to one of the following three arms: DPI-386 Nasal Gel + placebo patch, placebo nasal gel + placebo patch, or placebo nasal gel + TDS patch.

Treatment Day 1 will be conducted aboard an ocean-going vessel to obtain data in an operationally relevant real world environment immediately followed by Treatment Days 2 and 3 at a clinical site or one of its two satellite locations.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed and dated Informed Consent Form (ICF).
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 to 59 (inclusive).
4. At least two responses on the MSSQ must be "Sometimes" or "Frequently".
5. In good general health as evidenced by medical history with no recent history or current diagnosis of uncontrolled clinical problems as assessed by the Principal Investigator (PI) or qualified designee.
6. Ability to take intranasal medication and willingness to adhere to the study schedule and time constraints.
7. For females of child-bearing potential: willingness to provide a urine sample for the hCG pregnancy test. The test must be negative within seven days of the Treatment Day 1.
8. Agreement to adhere to the following lifestyle compliance considerations:

   * Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the three Treatment Days.
   * Abstain from alcohol for 24 hours prior to first dose of study medication and during the three Treatment Days.

Exclusion Criteria:

1. Pregnancy, lactation, or positive urine pregnancy test within seven days of Treatment Day 1.
2. Known allergic reactions to scopolamine or other anticholinergics.
3. Currently prescribed any of the following medication types and used within the specified washout periods below:

   * any form of scopolamine (including Transderm Scop®) (washout 5 days)
   * belladonna alkaloids (washout 2 weeks),
   * antihistamines (including meclizine) (washout 2 weeks),
   * tricyclic antidepressants (washout 2 weeks),
   * muscle relaxants (washout 4 days) and
   * nasal decongestants (washout 4 days)
4. Hospitalization or significant surgery requiring hospital admittance within the past six months.
5. Treatment with another investigational drug or other intervention within the past 30 days.
6. Having donated blood or plasma or suffered significant blood loss within the past 30 days.
7. Having any of the following medical conditions within the last two years or if any of the following medical conditions were experienced more than two years ago and are deemed clinically significant by the PI or qualified designee:

   * Significant gastrointestinal disorder, asthma, or seizure disorders.
   * History of cardiovascular disease.
   * History of vestibular disorders.
   * History of narrow-angle glaucoma.
   * History of urinary retention problems.
   * History of alcohol or drug abuse.
   * Nasal, nasal sinus, or nasal mucosa surgery.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2019-06-09 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects who developed motion sickness. | 8 hours
  Number of Subjects who developed motion sickness
Adverse Event (AE) Reporting of DPI-386 | 7 weeks
  Number of subjects with indicated AEs receiving DPI-386

SECONDARY OUTCOMES:
Severity of nausea as measured by the Visual Analog Scale (VAS) | During the 8 hour voyage on Treatment Day 1.
  VAS - Respondents specify their degree of nausea by indicating a point along a continuous 100 mm line between two end-points; left one is for "No nausea" and the right one for "Very severe nausea". Scoring is based on the length from left point and a higher score means more severe degree of nausea (Spinks & Wasiak, 2011).
Severity of motion sickness as measured by the Motion Sickness Assessment Questionnaire (MSAQ) over the treatment period. | During the 8 hour voyage on Treatment Day 1.
  MSAQ - The MSAQ was designed to measure motion sickness as a multi-dimensional construct, with the understanding that when an individual states they are experiencing motion sickness, it is unlikely a single symptom, but rather a complex set of symptoms, with varying levels of severity. Sixteen symptoms are listed, with symptoms differentiated along four dimensions: gastrointestinal, central, peripheral, and sopite-related. Each symptom is scored from 1 to 9 in severity and scores then calculated. All 16 items were collected from the general public instead of experts, allowing for a more accurate wording of the symptomology experienced by persons outside of physiological sciences. The MSAQ has been repeatedly validated and is strongly correlated with both the Pensacola Diagnostic index (r = 0.81, p < 0.001) and the Nausea Profile (r = 0.92, p < 0.001).
3. Cognition as measured by the Automated Neuropsychological Assessment Metrics (ANAM). | During all three Treatment Days.
  This battery consists of the ANAM CORE battery plus the Running Memory Continuous Performance Test (CPT).
Pharmacokinetic parameters of DPI-386 to be measured will include Maximum Observed Plasma Concentrations (Cmax) | On Treatment Days 2 -3, PK draws will occur at the following time points: -60, 30, 60, 90, 120, 180, 330, 390, 450, 480 and 600 minutes.
  Pharmacokinetics will be assessed by the amount of total free scopolamine at each time point blood is collected and plasma samples will be assayed for scopolamine using a fully validated LC/MS method.
Pharmacokinetic parameters of DPI-386 to be measured will include Time to Reach Maximum Observed Plasma Concentration (tmax). | On Treatment Days 2 -3, PK draws will occur at the following time points: -60, 30, 60, 90, 120, 180, 330, 390, 450, 480 and 600 minutes.
  Pharmacokinetics will be assessed by the amount of total free scopolamine at each time point blood is collected and plasma samples will be assayed for scopolamine using a fully validated LC/MS method.
Pharmacokinetic parameters of DPI-386 to be measured will include Area Under the Curve (AUC). | On Treatment Days 2 -3, PK draws will occur at the following time points: -60, 30, 60, 90, 120, 180, 330, 390, 450, 480 and 600 minutes.
  Pharmacokinetics will be assessed by the amount of total free scopolamine at each time point blood is collected and plasma samples will be assayed for scopolamine using a fully validated LC/MS method.

CONTACTS AND LOCATIONS:
Overall Officials: David R Helton, Study Director — Repurposed Therapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
Publication